CLINICAL TRIAL: NCT02884219
Title: Multi-center, Randomized Non-inferiority Trial of Early Treatment Versus Expectative Management of Patent Ductus Arteriosus in Preterm Infants (BeNeDuctus Trial - Belgium Netherlands Ductus Trial)
Brief Title: Early Treatment Versus Expectative Management of PDA in Preterm Infants
Acronym: BeNeDuctus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 843002622
Record Dates: First submitted 2016-04-01; First posted 2016-08-30 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2020-04

CONDITIONS: Patent Ductus Arteriosus
Keywords: Early treatment; Expectative treatment; Patent ductus arteriosus; Preterm
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Ibuprofen; Cyclooxygenase Inhibitors; Conservative Treatment; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Treatment with cyclooxygenase inhibitors (Active Comparator): Treatment of PDA that starts within the first 3 days of life using cyclooxygenase-inhibitors (Ibuprofen or Indomethacin)
  Interventions: Drug: Ibuprofen; Drug: Indomethacin
- Expectative Treatment (Sham Comparator): Expectative PDA management is characterized as 'watchful waiting'. No intervention is initiated with the intention to close a PDA.
  Interventions: Other: Expectative Management

INTERVENTIONS:
Drug: Ibuprofen — In the medical treatment (COXi) arm the intention is to close the ductus arteriosus.
  Other Names: Cyclooxygenase Inhibitor
  Arms: Early Treatment with cyclooxygenase inhibitors
Other: Expectative Management — Expectative PDA management is characterized as 'watchful waiting'. No intervention is initiated with the intention to close a PDA.
  Other Names: Conservative management
  Arms: Expectative Treatment
Drug: Indomethacin — In the medical treatment (COXi) arm the intention is to close the ductus arteriosus.
  Other Names: Cyclooxygenase Inhibitor
  Arms: Early Treatment with cyclooxygenase inhibitors

SUMMARY:
Much controversy exists about the optimal management of a patent ductus arteriosus (PDA) in preterm infants, especially in those born at a gestational age <28 weeks and/or a birth weight ≦1000 grams due to a lack of evidence for or against different approaches. A PDA has been associated with serious complications. However, a common finding is that medical and/or surgical treatment of a PDA seems not to reduce the risk of mortality or major morbidity. This might be related to the fact that a substantial portion of preterm infants are treated unnecessarily, because the ductus arteriosus (DA) might have closed spontaneously without any specific intervention. An expectative approach is gaining interest, although convincing evidence is still missing.

The objective of this study is to investigate whether in preterm infants <28 weeks' gestation with a PDA an expectative management is not inferior to early treatment with regard to the composite of mortality and/or necrotizing enterocolitis (NEC) and/or bronchopulmonary dysplasia (BPD) at a postmenstrual age of 36 weeks.

DETAILED DESCRIPTION:
After obtainment of informed consent the first echocardiographic evaluation is performed at a postnatal age of 24-72 hours. In absence of exclusion criteria patients will only be randomized when a PDA is present, the transductal diameter measures >1.5 mm and a blood flow pattern with a predominantly left-to-right shunt is observed. Randomization will assign the neonate to either the medical treatment (COXi) arm or the expectative PDA management arm.

It is essential that neonatal management is similar in both arms with the exception of the prescription of COX-inhibition and routine echocardiographic examination after a course of COXi in the medical treatment arm.

Medical treatment arm When the patient is allocated to the medical treatment arm COX-inhibition is prescribed and started as soon as possible, but no later than 3 hours after the echocardiogram.

The investigators prefer to use Ibuprofen (IBU) for COX-inhibition in this study. Aside from the above mentioned reasons the investigators are confronted with an actual lack of availability of indomethacin in most centers in the Netherlands and Belgium. However, Indomethacin (INDO) can be prescribed for medical ductal closure if this is preferred by a participating center.

The dosing schemes for IBU and INDO are according the local guidelines. For the first week of life the birth weight is used for calculation of the COXi dosage. After a postnatal age of 7 days the actual weight is used for dose calculation, except when the actual weight is still less than the birthweight.

The treatment described above is considered standard of care in many NICU's worldwide. It should be noted that there is no modification of the commonly advised usage of IBU in this study. There are reports that suggest that an high dose of IBU might be more effective in ductal closure in preterm infants, especially in those less than 27 weeks' gestation. However, in a systematic review one refrained from recommendations regarding high dose IBU because of the limited number of patients enrolled in studies.

The preferred route of administration of IBU is intravenously. However, this is at the disposal of the attending physician, since enteral administration appears at least as effective.

Echocardiographic reevaluation is performed at least 12 hours after the last (3rd) dose of the first COXi course. If the ductus arteriosus is found to be closed, no further analysis or treatment is needed regarding the ductus arteriosus. A ductus arteriosus is considered to be closed when it can't be visualized using color Doppler imaging or when the transductal diameter measures less than 0.5 mm.

When the ductus arteriosus hasn't closed, a second course of COX-inhibition is started at least 24 hours after the third dose of the first course. COXi dosages are similar to the first course.

Twelve to 24 hours after the last dose of the second course (6th gift) echocardiography is performed. If the ductus arteriosus is found to be closed, no further analysis or treatment is needed regarding the ductus arteriosus.

When the duct failed to close after two courses of COXi (6 doses in total) and the PDA is judged to be still hemodynamically significant, ductal ligation can be considered, only when the so-called 'ligation criteria' are met.

Expectative PDA management arm Patients randomized to the expectative management arm will not receive any COXi and PDA management in this group can be characterized as "watchful waiting". This is not a unique approach, since a restrictive approach towards a PDA is increasingly used in many centers worldwide without the observation of an increased risk of neonatal mortality and morbidity, such as severe chronic lung disease (CLD), intraventricular hemorrhage (IVH), NEC and retinopathy of prematurity (ROP).

It is essential that neonatal management is similar in both study arms with the exception of the prescription of COXi and echocardiography at the end of the drug course in the medical treatment arm. It is of the upmost importance that NO extra interventions are to be undertaken with the intention to conservatively prevent or treat a (suspected) PDA in the expectative arm, such as fluid restriction and diuretics for that reason. Moreover, it should be noted that there is insufficient evidence that fluid restriction and/or diuretics are of any benefit in patients with a (suspected) PDA.

When during the first week the attending physician is of the opinion that the patient is in danger, when it's deprived from treatment with COXi, open label treatment can only be considered when the 'open label criteria' are met.

ELIGIBILITY:
Inclusion Criteria:

* PDA diameter > 1.5 mm and ductal (predominantly) left-to-right shunt
* Signed informed consent obtained from parent(s) or representative(s)
* Gestational age < 28 completed weeks

Exclusion Criteria:

* Contraindication for administration of cyclooxygenase-inhibitors (COXi)
* Persistent pulmonary hypertension (ductal right-to-left shunt ≧33% of cardiac cycle)
* Congenital heart defect, other than PDA and/or patent foramen ovale (PFO)
* Life-threatening congenital defects
* Chromosomal abnormalities and/or congenital anomalies associated with abnormal neurodevelopmental outcome
* Use of COXi prior to randomization

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Composite of mortality, and/or NEC, and/or BPD | At a postmenstrual age of 36 completed weeks
  The primary outcome is the composite of mortality, and/or NEC (Bell stage ≥ IIa), and/or BPD, defined as the need for supplemental oxygen need, all at a postmenstrual age of 36 completed weeks.

SECONDARY OUTCOMES:
Short term sequelae of cardiovascular failure | Day 1 up to 3 months
  At the time of discharge the incidence of cardiovascular failure is calculated
Short term sequelae of adverse events | Day 1 up to 3 months
  At the time of discharge the number of all adverse events are calculated
Long-term neurodevelopmental consequences assessed with BSID-III-NL. | Assessed at an corrected age of 2 years
  All patients in this study will be included in the National Neonatal Follow Up Program and are therefore seen at a corrected age of 24 months. Their neurodevelopment is assessed with the Bayley Scales of Infant and Toddler Development, Third Dutch Edition (BSID-III-NL).

CONTACTS AND LOCATIONS:
Overall Officials: Willem P de Boode, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (13):
- Belgium (3):
  - University Hospital Antwerp, Antwerp
  - Hôpital Erasme - Clinique Universitaires de Bruxelles, Brussels
  - University Hospital Brussels, Brussels
- Netherlands (10):
  - Academic Medical Center, Amsterdam
  - Free University Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maatricht University Medical Center, Maastricht
  - Radboudumc Amalia Children's Hospital, Nijmegen
  - Erasmus Medical Center Rotterdam, Rotterdam
  - Wilhelmina Children's Hospital/UMCU, Utrecht
  - Maxima Medical Center, Veldhoven
  - Isala Kliniek Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available after an embargo period

REFERENCES:
- [Result] Hundscheid T, Onland W, Kooi EMW, Vijlbrief DC, de Vries WB, Dijkman KP, van Kaam AH, Villamor E, Kroon AA, Visser R, Mulder-de Tollenaer SM, De Bisschop B, Dijk PH, Avino D, Hocq C, Zecic A, Meeus M, de Baat T, Derriks F, Henriksen TB, Kyng KJ, Donders R, Nuytemans DHGM, Van Overmeire B, Mulder AL, de Boode WP; BeNeDuctus Trial Investigators. Expectant Management or Early Ibuprofen for Patent Ductus Arteriosus. N Engl J Med. 2023 Mar 16;388(11):980-990. doi: 10.1056/NEJMoa2207418. Epub 2022 Dec 6. PMID 36477458
- [Derived] Hundscheid T, Donders R, Onland W, Kooi EMW, Vijlbrief DC, de Vries WB, Nuytemans DHGM, van Overmeire B, Mulder AL, de Boode WP; BeNeDuctus trial study group. Multi-centre, randomised non-inferiority trial of early treatment versus expectant management of patent ductus arteriosus in preterm infants (the BeNeDuctus trial): statistical analysis plan. Trials. 2021 Sep 15;22(1):627. doi: 10.1186/s13063-021-05594-x. PMID 34526095
- [Derived] Hundscheid T, Onland W, van Overmeire B, Dijk P, van Kaam AHLC, Dijkman KP, Kooi EMW, Villamor E, Kroon AA, Visser R, Vijlbrief DC, de Tollenaer SM, Cools F, van Laere D, Johansson AB, Hocq C, Zecic A, Adang E, Donders R, de Vries W, van Heijst AFJ, de Boode WP. Early treatment versus expectative management of patent ductus arteriosus in preterm infants: a multicentre, randomised, non-inferiority trial in Europe (BeNeDuctus trial). BMC Pediatr. 2018 Aug 4;18(1):262. doi: 10.1186/s12887-018-1215-7. PMID 30077184
- See also: Website BeNeDuctus Trial — https://neonatology.eu/studies/beneductus